CLINICAL TRIAL: NCT06694545
Title: Role of Intravenous Magnesium Sulphate and Caffeine in Neonates with Hypoxic Ischemic Encephalopathy (HIE) in a Assiut University Hospital of Children
Brief Title: Neonates with Hypoxic Ischemic Encephalopathy (HIE)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Malak Zaki Malak, 71515,Assiut, Assiut University
Other Study IDs: Hypoxic IschemicEncephalopathy
Record Dates: First submitted 2024-09-06; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hypoxic Ischemic Encephalopathy (HIE)
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Assessment of the potential neuroprotective effect of magnesium sulphate and caffeine in treating asphyxiated newborns and improvement of the neurological outcome of Hypoxic Ischemic Encephalopathy in Assiut university hospital of Children

DETAILED DESCRIPTION:
Encephalopathy in neonates is broadly defined as brain dysfunction in a newborn manifesting as alteration in mental status and abnormal neurologic examination. Neonatal encephalopathy (NE) may result from acute or chronic hypoxic-ischemic injury, brain malformations, vascular injuries (including stroke), inborn errors of metabolism, and other causes. Hypoxic-ischemic encephalopathy (HIE) is a specific diagnosis and applies only when a neonate has encephalopathy that is known or highly suspected to be due to a hypoxic-ischemic event.

Perinatal asphyxia is a condition where hypoxaemia and acidosis are present in the fetus or the newborn infants. It is a failure newborn to initiate spontaneous, sustained, and vigorous respiration effort at birth. It is also defined as a failure to initiate spontaneous respirations and/or a 5-minute Apgar score of less than 7: the most commonly used indicator in the identification of birth asphyxia in resource limited settings . About 20% - 30% of asphyxiated newborns who develop hypoxic ischemic encephalopathy (HIE) die during the neonatal period, and one third to one half of survivors are left with cerebral palsy and mental retardation . Survivors present with several short and long term morbidities, including: seizure disorders, tone abnormalities, feeding difficulties, delayed developmental milestones, learning difficulties, cerebral palsy and mental retardation. The frequency of severe perinatal asphyxia complications, hypoxic ischemic encephalopathy (HIE) and incidence of up to 26.5/1000 live births is unacceptably high despite advances in perinatal care . Encephalopathy occurs in 50% to 60% of patients with severe perinatal asphyxia. Among patients with moderate HIE, 10% to 20% die, and 30% to 40% develop neurodevelopmental disorders, whereas 50% of patients with severe HIE die and almost all survivors develop neurodevelopmental deficits Neuro-science research has revealed our understanding of the mechanisms by perinatal asphyxia neuronal damage and adverse consequences. Asphyxia leads to two types of cerebral injuries: the primary neuronal injury that occurs at the time of hypoxic-ischemic insults and the secondary cerebral injury that occurs over hours to days after accumulation of excessive intra-neuronal calcium through stimulation of the excitatory N-methyl-D-aspartate (NMDA) glutamate receptors, which triggers apoptosis of the affected neurons . Magnesium is a naturally occurring NMDA receptor antagonist that blocks neuronal influx of calcium within the ion channels. This block is voltage-dependent and is overcome during axonal depolarization that occurs in hypoxic-ischemic insults. If the extra-cellular magnesium concentration is increased, this blockade can be restored. Magnesium sulphate may also have direct actions on mitochondrial activity, anticonvulsant properties and hemodynamic effects by increasing cerebral blood flow. Some data also suggest that MgSO4 may serve an anti-apoptotic role and prevent neuronal cell loss .

Clinical studies have shown that caffeine also has neuroprotective effects in premature infants by alleviating hypoxia induced white matter damage, and improving ventilation function and brain self-regulation In addition, caffeine has been shown to reduce the apoptosis of developing brain neurons, ventricular enlargement, and white matter loss caused by hypoxia.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with suspected perinatal asphyxia APGAR score < 3 at 5 min.
2. Neonates whose mother did not receive MgSO4 or caffeine

Exclusion Criteria:

1. Neonates with Apgar's score > 3 at 5 min
2. Neonates with congenital malformations
3. Neonates whose mother had general anasthesia

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with Hypoxic Ischemic Encephalopathy (HIE) .Encephalopathy in neonates is broadly defined brain dysfunction in a newborn manifesting as alteration in mental status and abnormal neurologic examination. Neonatal encephalopathy (NE) may result from acute or chronic hypoxic-ischemic injury, brain malformations, vascular injuries (including stroke), inborn errors of metabolism, and other causes. Hypoxic-ischemic encephalopathy (HIE) is a specific diagnosis and applies only when a neonate has encephalopathy that is known or highly suspected to be due to a hypoxic-ischemic event.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the potential neuroprotective effect of magnesium sulphate and caffeine in improvement of the neurological outcome of hypoxic ischemic encephalopathy in Assuit university hospital. | Baseline
  Assesment of neuroprotective effect of magnesium sulphate and caffeine by :
  1. Determine the benefit of magnesium sulphate and caffeine on perinatal asphyxia.
  2. Determine the effect of magnesium sulphate and caffeine on neurological outcome in severe perinatal Asphyxia.
  3. Determine the effect of magnesium sulphate and caffeine on reduction of duration of Admission/hospitalization.

REFERENCES:
- [Background] Azra Haider B, Bhutta ZA. Birth asphyxia in developing countries: current status and public health implications. Curr Probl Pediatr Adolesc Health Care. 2006 May-Jun;36(5):178-88. doi: 10.1016/j.cppeds.2005.11.002. No abstract available. PMID 16631096
- [Background] Chalak L, Ferriero DM, Gressens P, Molloy E, Bearer C. A 20 years conundrum of neonatal encephalopathy and hypoxic ischemic encephalopathy: are we closer to a consensus guideline? Pediatr Res. 2019 Nov;86(5):548-549. doi: 10.1038/s41390-019-0547-9. Epub 2019 Aug 26. No abstract available. PMID 31450231
- [Background] Volpe JJ. Neonatal encephalopathy: an inadequate term for hypoxic-ischemic encephalopathy. Ann Neurol. 2012 Aug;72(2):156-66. doi: 10.1002/ana.23647. PMID 22926849